CLINICAL TRIAL: NCT02321904
Title: Corneal Confocal Microscopy to Detect Diabetic Neuropathy in Children
Acronym: CCM
Status: Completed | Type: Observational
Sponsor: University of Calgary (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Dr. Danièle Pacaud, Associate Professor, University of Calgary
Other Study IDs: E-21944
Record Dates: First submitted 2013-06-17; First posted 2014-12-22 (Estimated); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Type 1 Diabetes; Neuropathy; Retinopathy
Keywords: Confocal microscopy; Cornea; Neuropathy; Detection; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Retinal Diseases; Corneal Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic cases: Children with Type 1 Diabetes 8 to 18 years old followed at the Alberta Children's Hospital Diabetes Clinic with duration of diabetes for at least 5 years will undergo Corneal Confocal Microscopy, Nerve Conduction Studies, Quantitative sensory testing, Neuropathy Symptom Scoring and Clinical nerve examinations.
  Interventions: Procedure: Corneal Confocal Microscopy; Procedure: Nerve Conduction Studies; Procedure: Quantitative sensory testing; Procedure: Neuropathy Symptom Score; Procedure: Clinical nerve examination
- Normal controls: Healthy children aged 8 to 18 years will undergo Corneal Confocal Microscopy, Nerve Conduction Studies, Quantitative sensory testing, Neuropathy Symptom Scoring and Clinical nerve examinations.
  Interventions: Procedure: Corneal Confocal Microscopy; Procedure: Nerve Conduction Studies; Procedure: Quantitative sensory testing; Procedure: Neuropathy Symptom Score; Procedure: Clinical nerve examination

INTERVENTIONS:
Procedure: Corneal Confocal Microscopy — Close-up pictures of the front part of the eye (the cornea)
Procedure: Nerve Conduction Studies — The following assessments will be made: a) amplitude of nerve action potential (μV) and conduction velocity (m/s) of the sural sensory nerve by antidromic stimulation; b) motor nerve conduction velocity (m/s), maximum M-wave amplitude (mV) and motor nerve distal latency (ms) of the peroneal motor nerve; and c) tibial nerve conduction study will also be obtained if tolerated.
Procedure: Quantitative sensory testing — Standardized vibratory and thermal stimulation levels applied to the subject's non-dominant big toe.
Procedure: Neuropathy Symptom Score — A list of 18 motor, sensory and autonomic symptoms encountered in a diabetic patients with neuropathy obtained by interview.
Procedure: Clinical nerve examination — Summated score of the lower extremities. Neurological examination assessing muscle strength, knee and ankle reflexes, sensation in the great toes will be evaluated for light touch-pressure, temperature, pin-prick, vibratory sense and joint position sense.

SUMMARY:
The overall aim of this study is to confirm the utility of corneal confocal microscopy (CCM) as a new technique to rapidly and non-invasively assess diabetic neuropathy (DN) in children. This study will be divided into two phases: Phase 1 will be a cross-sectional study of children with type 1 diabetes and normal controls, while phase 2 will be a longitudinal assessment of a subgroup of children with type 1 diabetes recruited during Phase 1.

DETAILED DESCRIPTION:
In phase 1: To compare corneal nerve density (CND), length (CNL), and branching (CBD) by CCM between

1. children with type 1 diabetes for 5 years or more to children without diabetes;
2. children with type 1 diabetes with and without evidence of diabetic neuropathy;
3. to examine the relationship between CND, CNL & CBD and known risk factors of diabetic neuropathy

In phase 2:

1. to examine for changes in corneal nerve morphology two years after the initial CCM exam.
2. to describe the evolution of diabetic neuropathy based on clinical symptoms, neurological deficits, and other tests of nerve dysfunction.
3. to assess if changes in corneal nerve morphology correlate with changes in nerve conduction velocity and autonomic testing.
4. To examine the risk factors associated with progression of diabetic neuropathy in our pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* CASES: Children with Type 1 Diabetes 8 to 18 years old followed at the Alberta Children's Hospital Diabetes Clinic with a duration of diabetes of at least 5 years.
* CONTROLS: Healthy children aged 8 to 18 years.

Exclusion Criteria:

* Patients with known history of corneal abnormality, trauma, or surgery
* Any other cause of neuropathy
* Individuals with uncontrolled hypothyroidism
* Individuals with celiac disease
* Other serious chronic illnesses besides diabetes
* Inability to cooperate with testing
* Families unwilling to provide written informed consent

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Cases: Children seen at the Alberta Children's Hospital Diabetes Clinic in Calgary Controls: 8-18 year old healthy children
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2008-06; Primary Completion 2014-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
The utility of corneal confocal microscopy to assess diabetic neuropathy in children. | 2 years
  To confirm the utility of corneal confocal microscopy (CCM) as a new technique to rapidly assess diabetic neuropathy (DN) in children. This non-invasive eye imaging method may be a superior alternative to traditional nerve conduction studies.
  This study will be divided into two phases: Phase 1 will be a cross-sectional study of children with Type 1 Diabetes (T1D) and normal controls, while phase 2 will be a longitudinal assessment of a subgroup of T1D children recruited during Phase 1.

SECONDARY OUTCOMES:
Corneal nerve density (CND) by CCM | Single time point
  To compare corneal nerve density (CND) between
  1. children with T1D for 5 years or more to children without diabetes;
  2. children with T1D with and without evidence of DN;
  3. to examine the relationship between CND, CNL & CBD and known risk factors of DN
Changes in corneal nerve morphology two years after the initial CCM exam. | 2 years
  In phase 2 : 1) to examine for changes in corneal nerve morphology two years after the initial CCM exam.
  2) to describe the evolution of DN in based on clinical symptoms, neurological deficits, and other tests of nerve dysfunction.
  3) to assess if changes in corneal nerve morphology correlate with changes in nerve conduction velocity and autonomic testing. 4) To examine the risk factors associated with progression of DN in our pediatric population.
Corneal nerve length (CNL) by CCM. | Single time point
  To compare corneal nerve length (CNL), by CCM between
  1. children with T1D for 5 years or more to children without diabetes;
  2. children with T1D with and without evidence of DN;
  3. to examine the relationship between CND, CNL & CBD and known risk factors of DN
Corneal nerve branching density (CBD) by CCM | Single time point
  To compare corneal nerve branching density (CBD) by CCM between
  1. children with T1D for 5 years or more to children without diabetes;
  2. children with T1D with and without evidence of DN;
  3. to examine the relationship between CND, CNL & CBD and known risk factors of DN

CONTACTS AND LOCATIONS:
Overall Officials: Danièle Pacaud, Md, FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Alberta Children's Hospital, Calgary, Alberta, Canada